CLINICAL TRIAL: NCT00352508
Title: The Dietary Intervention in e-Shopping Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: Diet2006
Record Dates: First submitted 2006-03-19; First posted 2006-07-14 (Estimated); Last update posted 2006-07-14 (Estimated); Status verified 2006-03

CONDITIONS: Behaviour
Keywords: Internet, dietary advice, saturated fat
MeSH Terms: conditions — Behavior | interventions — Nutrition Assessment

INTERVENTIONS:
Behavioral: Dietary advice

SUMMARY:
The supermarket industry now services many customers through online food shopping over the Internet. The Internet shopping process offers a novel opportunity for the modification of dietary patterns. The aim of this study was to evaluate the effects on consumers' purchases of saturated fat of a fully automated computerised system that provided real-time, personally tailored advice recommending foods lower in saturated fat.

DETAILED DESCRIPTION:
Objective The supermarket industry now services many customers through online food shopping over the Internet. The Internet shopping process offers a novel opportunity for the modification of dietary patterns. The aim of this study was to evaluate the effects on consumers' purchases of saturated fat of a fully automated computerised system that provided real-time, personally tailored advice recommending foods lower in saturated fat.

Design Blinded, randomized controlled trial.

Setting & Participants Consumers using a commercial on-line Internet shopping site between February and June 2004.

Intervention Individuals assigned to intervention received fully automated individually tailored advice that recommended specific switches from selected products higher in saturated fat to alternate similar products lower in saturated fat. Participants assigned to control received general non-specific advice about how to eat a diet lower in saturated fat.

Outcome measure The percent of food purchased that was saturated fat. Results There were 497 randomised participants, mean age 40 each shopping for an average of about 3 people. The amount of saturated fat in the foods purchased by the intervention group was 0.66% lower (95% confidence interval 0.48-0.84, p<0.0001) than in the control group. The effects of the intervention were sustained over time and there was no difference in the average cost of the food bought by each group.

Conclusions Fully automated, personally tailored dietary advice offered to customers doing Internet shopping can bring about changes in food purchasing habits that are likely to have significant public health implications. Because implementation is simple to initiate and maintain this strategy would likely be highly cost-effective.

ELIGIBILITY:
Inclusion Criteria:

- Consumers using a commercial on-line Internet shopping site between February and June 2004.

Exclusion Criteria:

Children, non-internet shoppers

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2004-09; Study Completion 2004-12

PRIMARY OUTCOMES:
The percent of food purchased that was saturated fat.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Neal, PhD, Principal Investigator — The George Institute
Locations (1):
- The George Institute, Sydney, New South Wales, Australia